CLINICAL TRIAL: NCT07008625
Title: The Effect of Virtual Reality Application on Anxiety and Milk Quantity in Mothers Who Milk Their Babies by Milking
Brief Title: the Effect of Virtual Reality Glasses on Women Who Milk Their Babies by Milking
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Collaborators: Zeynep Kamil Maternity and Pediatric Research and Training Hospital (Other)
Responsible Party: Principal Investigator, Zümrüt Bingin, associate professor, Marmara University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MU-SBF-ZB-01
Record Dates: First submitted 2025-05-29; First posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-05

CONDITIONS: Human Milk, Breast Milk
Keywords: Breast milk, milking, newborn, virtual reality glasses

STUDY DESIGN:
Intervention Model Description: It is a randomized controlled experimental research type.
Who Masked: Investigator
Masking Description: virtual reality glasses will be applied to the experimental group that was blinded, and routine clinical care will be given to the control group that was blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): virtual reality glasses will be applied
  Interventions: Device: virtual reality glasses
- control group (Active Comparator): only routin clinical care will be applied
  Interventions: Behavioral: routine care

INTERVENTIONS:
Device: virtual reality glasses — Experimental Group (Those who applied virtual reality glasses):
  1.Stage: The mothers who will be included in the experimental-application group will first be informed about the study and the "Informed Volunteer Consent Form" will be filled out. Then to mothers (breast milk, methods of milking, etc.) information will be provided about. Before milking, the "Personal Information Form", the "Status Anxiety Scale", the "Inadequate Milk Perception Scale" will be applied. After the application of the forms and scales to be used in the study 1.the milking process will be performed (If milking is to be done with a milking machine, the device used will be "Babyvacc Model TBM3100".) and the amount of milk milked will be measured (in a plastic 150 ml sized bottle contained in the Milkvacc breast milk milking and storage kit belonging to Ankalaps Company), and attention will be paid to the inclusion of mothers who have never been able to breastfeed for medical reasons in the study.
  Mothers in the
  Arms: experimental group
Behavioral: routine care — 1.Stage: The mothers who will be included in the control group will first be informed about the study and the "Informed Volunteer Consent Form" will be filled out. Then to mothers (breast milk, methods of milking, etc.) information will be provided about. Before milking, the "Personal Information Form", the "Status Anxiety Scale", the "Inadequate Milk Perception Scale" will be applied. After the application of the forms and scales to be used in the study, 1.the milking process will be performed (If milking is to be done with a milking machine, the device used will be "Babyvacc Model TBM3100".) and the amount of milk milked will be measured (in a plastic 150 ml sized bottle contained in the Milkvacc breast milk milking and storage kit belonging to Ankalaps Company), and attention will be paid to the inclusion of mothers who have never been able to breastfeed for medical reasons in the study.
  Mothers in the control group were given 1 during the waiting for the next milking time. and 2. r
  Arms: control group

SUMMARY:
The research was conducted at the Istanbul Zeynep Kamil Women's And Children's Diseases Education And Research Hospital's Maternity Service between the dates of June 15 and December 31, 2025. It is a randomized controlled experimental research. The data consist of a total of 32 primiparous mothers whose baby was hospitalized in the neonatal intensive care unit who met the criteria for inclusion in the study. Mothers were divided into groups (16 experiments, 16 controls) by randomization method. The data of the research were collected using the Personal Information Form, the Status Anxiety Scale and the Inadequate Milk Perception Scale after obtaining the permission of the ethics committee and the institution. Virtual reality glasses were applied to the mothers in the experimental group. Only routine clinical care was applied to the mothers in the control group.

DETAILED DESCRIPTION:
Type of Research: It is a randomized controlled experimental research type.February Decembers/Sample of the Research: The research will be conducted between 3 February 2025-31 December 2025 after obtaining the approval of the ethics committee and the authorizations of the institution.

February December 3, 2025-31, 2025, SBU Zeynep Kamil Women's and Children's Diseases Training and Research Hospital Dec. 3, 2025, the universe of the research will be composed of primiparous mothers whose baby is hospitalized in the neonatal unit. Primiparous mothers (a total of 32 mothers) who participated wholeheartedly in the study will constitute the sample.

Working Group Power analysis was performed to determine the number of people to be included in the research. The strength of the test was calculated using the G*Power 3.1 program. As a similar research in the relevant literature, the effect size of the change in the amount of breast milk was calculated as 1.354 in the study conducted by Herlina et al. (2022). In order to exceed the 99% value in determining the strength of the study, it is necessary to reach 26 people, including 13 people in groups with a significance level of 5% and an effect size of 1,354(df=41; t=1,683). In the research, it was aimed to reach a total of 32 people, including 16 people in groups, taking into account the high strength of the test and the losses.

Statistical Analysis of the Data The data obtained in the research will be analyzed using the Statistical Package for Social Sciences (SPSS) for Windows 22.0 program. The Kolmogorov Smirnov Test will be used to determine whether the research data are distributed normally. According to the Kolmogorov Smirnov Test, if p>0.05, the distribution is determined to be normal. However, if p<0.05, it is determined that the distribution is not normal and the Skewness and Kurtosis values of the data are checked. If the Skewness and Kurtosis values are between +2 and -2, it is assumed that the variable shows a normal distribution (George, Dec and Mallery, 2010). The homogeneity of the descriptive characteristics between the groups will be tested by chi-square analysis.Dec. For the difference between the averages of two independent groups, the data will be evaluated using the t-test if they are Decently distributed, and the Mann-Whitney U test if the data are not decently distributed. Changes in measurements within the group if the data are distributed normally, repeated measurements will be analyzed by Anova test, and if the data are not distributed normally, Friedman test.

The Hypotheses of the Research H1. Virtual reality application is effective in increasing the amount of breast milk.

H2. Virtual reality application is not effective in increasing the amount of breast milk.

H3. Virtual reality application is effective in reducing mother's anxiety. H4. The virtual reality application is not effective in reducing the anxiety of the mother.

Collection of Data and Data Collection Tools After explaining that the purpose of the research and all kinds of information about them will be kept confidential to primiparous mothers who are hospitalized at SBU Zeynep Kamil Women's and Pediatrics Training and Research Hospital, whose babies receive care in the neonatal intensive care unit and meet the criteria for admission to the research, the Personal Information Form, the Status Anxiety Scale and the Inadequate Milk Perception Scale will be completed by the researchers using the face-to-face interview technique by having those who volunteer to participate sign an Informed Consent Form. The data collection time will take about 15-20 minutes.

* Personal Information Form: According to the relevant literature information provided by the researchers (Sari Ozturk and Demir, 2023; Ferraz Dos Santos et al., 2020) developed (Personal Information Form socio-demographic variables belonging to mothers (age, education level, income level, etc.) obstetric characteristics (pregnancy, miscarriage, number and shape of birth, etc.) consists of 33 questions related to breastfeeding and anxiety.
* State Anxiety Scale: The state-continuous anxiety scale is a self-assessment questionnaire consisting of short statements. It has been adapted to Turkish by Öner and Le Compte. In this study, only the State Anxiety subscale was used. The reason for this is that the Situational Anxiety Scale describes how an individual feels at a certain moment and under certain conditions, and includes a response taking into account their feelings about the situation they are in, Cronbach's Alpha internal consistency coefficient for the situational anxiety scale was found to be between 0.94 and 0.96 in reliability analyses. Dec. The state anxiety scale consists of a scale consisting of a total of twenty items. There is no time limit for responding to the scale. The emotions or behaviors expressed in the items of the state anxiety scale are answered by marking one of the following styles according to the degree of severity of such experiences: (1) none, (2) a little, (3) a lot, (4) completely. There are two types of expressions in the scale. We can call these direct or flat and inverted expressions. Direct expressions express negative emotions, while reversed expressions express positive emotions. When scoring these second types of expressions, those with a weight of 1 turn into 4, and those with a weight of 4 turn into 1. Responses with a value of 4 in direct statements indicate that anxiety is high. The reversed expressions are also; answers with a value of 1 indicate high anxiety, those with a value of 4 indicate low anxiety. The expression "I am restless" can be shown directly, and the expression "I Feel Calm" can also be shown as examples of reversed expressions. In this case, if 1 weighted option is selected for the expression "I am restless", these responses reflect high anxiety. There are ten reversed expressions in the Situational Anxiety Scale. These Are; 1, 2, 5, 8, 10, 11, 15, 16, 19 and they are the 20th articles. The total score of the direct and reversed expressions is calculated. From the total score obtained for direct expressions, the total score of reversed expressions is subtracted. A previously determined invariant value is added to this number. For the Status Anxiety Scale, this value is 50. In addition, this scale can score between 20-80 saras and one point above the standard deviation has been accepted as a cut-off point (Oner and Le Compte 1985).
* Inadequate Milk Perception Scale: Inadequate Milk Perception Scale The scale developed by McCarter-Spaulding and Kearney in 2001 consists of 6 questions to determine the inadequate perception of breast milk. The first question that questions whether the mother perceives her milk adequately is in the form of "yes" or "no". The other 5 questions are aimed at measuring the perception of milk Deciency and are scored between 0-10. "0" indicates that milk is completely inadequately perceived, "10" indicates that milk is completely adequately perceived. The scale is scored between 0-50 Dec. A high score indicates that the competence perception of milk has increased. The Cronbach α value was determined as 0.81 in the original of the scale (McCarter-Spaulding & Kearney, 2001). The validity reliability of the scale in Turkish was made by Gökçeoğlu and Küçükoğlu and the Cronbach α value of the study was found to be 0.82 (Gökçeoğlu, 2014).
* Virtual reality glasses (Game-Based) application: The content in the section "Methods of Milking" contained in the General Directorate of Public Health (HSGM) Breastfeeding Counseling Practitioner Book (2018) will be taken into account when determining the methods of breastfeeding that will be designed in the game in the research (HSGM, 2018). Since the easiest methods of milking are machine and manual milking methods, one of these methods will be selected as a milking method. Virtual reality application will be made to the experimental group and mothers will be informed about the method. Mothers who will apply the virtual reality glasses will be asked to choose any of 4 different types of videos and visuals from the visuals and videos designed for mothers to watch "during waiting for the milking time". The researcher, in accordance with the mother's request, will open the video or image determined by the mother while she is waiting for the milking time and help her watch it. He will be provided to watch videos and visuals at 1 hour intervals and for 15 minutes until the December milking time arrives.

The duration and frequency of watching all the designed videos and images will be determined as an average of 15 minutes according to the time of milking and filling the breasts with milk again.

10.6.2 Collection of Data

Experimental Group (Those who applied virtual reality glasses):

1. Stage: The mothers who will be included in the experimental-application group will first be informed about the study and the "Informed Volunteer Consent Form" will be filled out. Then to mothers (breast milk, methods of milking, etc.) information will be provided about. Before milking, the "Personal Information Form", the "Status Anxiety Scale", the "Inadequate Milk Perception Scale" will be applied. After the application of the forms and scales to be used in the study, 1.the milking process will be performed (If milking is to be done with a milking machine, the device used will be "Babyvacc Model TBM3100".) and the amount of milk milked will be measured (in a plastic 150 ml sized bottle contained in the Milkvacc breast milk milking and storage kit belonging to Ankalaps Company), and attention will be paid to the inclusion of mothers who have never been able to breastfeed for medical reasons in the study.

   Mothers in the experimental group will be told about the use of virtual reality glasses (SG) while waiting for the next milking time, and the first 1. Per hour and 2.SG will be applied per hour (1. Practice- 15 min), (2. practice-15 min). 2.2 for a period of 15-20 minutes at the end of the hour. the milking process will be performed.
2. Stage: After the milking process is completed, the "State Anxiety Scale" and the "Insufficient Milk Perception Scale" will be applied for the second time in the research.

Control Group (Those who underwent routine maintenance):

1. Stage: The mothers who will be included in the control group will first be informed about the study and the "Informed Volunteer Consent Form" will be filled out. Then to mothers (breast milk, methods of milking, etc.) information will be provided about. Before milking, the "Personal Information Form", the "Status Anxiety Scale", the "Inadequate Milk Perception Scale" will be applied. After the application of the forms and scales to be used in the study, 1.the milking process will be performed (If milking is to be done with a milking machine, the device used will be "Babyvacc Model TBM3100".) and the amount of milk milked will be measured (in a plastic 150 ml sized bottle contained in the Milkvacc breast milk milking and storage kit belonging to Ankalaps Company), and attention will be paid to the inclusion of mothers who have never been able to breastfeed for medical reasons in the study.

   Mothers in the control group were given 1 during the waiting for the next milking time. and 2. routine information will be provided during milking per hour and questions will be answered. 2.2 for a period of 15-20 minutes at the end of the hour. the milking process will be performed.
2. Stage: After the milking process is completed, the "State Anxiety Scale" used in the research and the "Insufficient Milk Perception Scale"will be applied for the second time. After that, information will be given to the mothers in this group about the application of virtual reality.

ELIGIBILITY:
Inclusion Criteria:

* • those between the ages of 18-35 December

  * Who is at least the first school graduate
  * Who can speak and understand Turkish
  * who gives birth to a single term at 37-42 weeks of pregnancy

    * The primiparous one
    * Who gives vaginal birth
  * Without any risk related to pregnancy and childbirth
  * The baby is in the neonatal intensive care unit
  * Giving milk to your baby by milking
  * Without any chronic systemic diseases

    * End of birth 1-4. what happened between the Dec
    * Mothers who volunteer to participate in the study and approve the consent document will be accepted to the study.

Exclusion Criteria:

* • With the loss of a baby during the study phase

  * Those who do not want to participate in the study or who voluntarily participated in the study but later gave up will be excluded from the study.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — only female
Enrollment: 32 (Estimated)
Dates: Start 2025-05-27 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Personal Information Form | 2 weeks
  In accordance with the relevant literature information provided by the researchers (Sari Ozturk and Demir, 2023; Ferraz Dos Santos et al., 2020) developed (Personal Information Form socio-demographic variables belonging to mothers (age, education level, income level, etc.) obstetric characteristics (pregnancy, miscarriage, number and shape of birth, etc.) consists of 33 questions related to breastfeeding and anxiety.
The Status Anxiety Scale | 2 weeks
  The status-continuous anxiety scale is a self-assessment questionnaire consisting of short statements. It has been adapted to Turkish by Öner and Le Compte. In this study, only the State Anxiety subscale was used. The reason for this is that the Situational Anxiety Scale describes how an individual feels at a certain moment and under certain conditions, and includes a response taking into account their feelings about the situation they are in, Cronbach's Alpha internal consistency coefficient for the situational anxiety scale was found to be between 0.94 and 0.96 in reliability analyses. Dec. The state anxiety scale consists of a scale consisting of a total of twenty items. There is no time limit for responding to the scale. The emotions or behaviors expressed in the items of the state anxiety scale are answered by marking one of the following styles according to the degree of severity of such experiences: (1) none, (2) a little, (3) a lot, (4) completely.
Inadequate Milk Perception Scale | 2 weeks
  Inadequate Milk Perception Scale Developed by McCarter-Spaulding and Kearney in 2001, the scale consists of 6 questions to determine the inadequate perception of breast milk. The first question that questions whether the mother perceives her milk adequately is in the form of "yes" or "no". The other 5 questions are aimed at measuring the perception of milk Deciency and are scored between 0-10. "0" indicates that milk is completely inadequately perceived, "10" indicates that milk is completely adequately perceived. The scale is scored between 0-50 Dec. A high score indicates that the competence perception of milk has increased. The Cronbach α value was determined as 0.81 in the original of the scale (McCarter-Spaulding & Kearney, 2001). The validity reliability of the scale in Turkish was made by Gökçeoğlu and Küçükoğlu and the Cronbach α value of the study was found to be 0.82 (Gökçeoğlu, 2014).

IPD SHARING:
Plan to Share IPD: No
I'm not sure to share my research.

REFERENCES:
- [Background] Karimi M, Haghighat M, Dialameh Z, Tahmasbi L, Parand S, Bardestani M. Breastfeeding as a Protective Effect Against Childhood Leukemia and Lymphoma. Iran Red Crescent Med J. 2016 Feb 13;18(9):e29771. doi: 10.5812/ircmj.29771. eCollection 2016 Sep. PMID 28144455
- [Background] Joshi A, Amadi C, Meza J, Aguire T, Wilhelm S. Evaluation of a computer-based bilingual breastfeeding educational program on breastfeeding knowledge, self-efficacy and intent to breastfeed among rural Hispanic women. Int J Med Inform. 2016 Jul;91:10-9. doi: 10.1016/j.ijmedinf.2016.04.001. Epub 2016 Apr 2. PMID 27185505
- [Background] Herlina, N., Ekowati, E., Fratidhina, Y., Nugroho, W., Agustina, I., & Aticeh, A. (2022). Virtual Reality (VR) Glasses for Oxytocin Relaxation Therapy to Increase Breast Milk Production of Postpartum Mothers. Jurnal Midpro. https://doi.org/10.30736/md.v14i1.418.
- [Background] Ferraz Dos Santos L, Borges RF, de Azambuja DA. Telehealth and Breastfeeding: An Integrative Review. Telemed J E Health. 2020 Jul;26(7):837-846. doi: 10.1089/tmj.2019.0073. Epub 2019 Oct 18. PMID 31633467
- [Background] Elgzar WT, Al-Thubaity DD, Alshahrani MA, Essa RM, Ibrahim HA. The Relationship between Maternal Ideation and Exclusive Breastfeeding Practice among Saudi Nursing Mothers: A Cross-Sectional Study. Nutrients. 2023 Mar 31;15(7):1719. doi: 10.3390/nu15071719. PMID 37049559
- [Background] Dantas DC, Goes FGB, Santos ASTD, Silva ACSSD, Silva MDA, Silva LFD. Production and validation of educational video to encourage breastfeeding. Rev Gaucha Enferm. 2022 Aug 15;43:e20210247. doi: 10.1590/1983-1447.2022.20210247.en. eCollection 2022. English, Portuguese. PMID 35976384
- [Background] Chen FQ, Leng YF, Ge JF, Wang DW, Li C, Chen B, Sun ZL. Effectiveness of Virtual Reality in Nursing Education: Meta-Analysis. J Med Internet Res. 2020 Sep 15;22(9):e18290. doi: 10.2196/18290. PMID 32930664
- [Background] Armstrong M, Lun J, Groner JI, Thakkar RK, Fabia R, Noffsinger D, Ni A, Keesari R, Xiang H. Mobile phone virtual reality game for pediatric home burn dressing pain management: a randomized feasibility clinical trial. Pilot Feasibility Stud. 2022 Aug 18;8(1):186. doi: 10.1186/s40814-022-01150-9. PMID 35982492